CLINICAL TRIAL: NCT03354858
Title: Oocyte Recovery Rate Following Follicular Flushing Versus Direct Aspiration in Women Undergoing IVF
Brief Title: Follicular Flushing Versus Direct Aspiration
Status: Completed | Type: Observational
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Other Study IDs: Follicular flushing
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Infertility
Keywords: follicle flushing; direct follicle aspiration; fertilization rate; maturation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Follicular flushing: One ovary will be aspirated using follicular flushing (up to 5 times per follicle).
  Interventions: Procedure: Follicular flushing
- No flushing: One ovary will be aspirated using direct aspiration (no flushing).

INTERVENTIONS:
Procedure: Follicular flushing — Repeated follicle flushing up to 5 times using a double lumen needle for oocyte recovery
  Groups: Follicular flushing

SUMMARY:
The purpose of this study is to investigate the impact of follicular flushing on the oocyte recovery rate, oocyte maturity, fertilization rate, and embryo development and utilization as compared to direct aspiration (no flushing) in women undergoing IVF treatment

DETAILED DESCRIPTION:
This will be a prospective observational paired study on the effect of follicular flushing oocyte recovery rate, oocyte maturity, fertilization rate, and embryo development and utilization as compared to direct aspiration (no flushing) in women undergoing IVF treatment.

In each woman enrolled, one ovary (right or left) will be randomly assigned to be aspirated with either follicular flushing or direct aspiration without flushing. The primary endpoint will be oocyte recovery rate (oocytes retrieved per follicle aspirated). Secondary outcomes will be oocyte maturity, fertilization rate, and embryo development and utilization. Pregnancy rates will be reported as a surrogate outcome.

TRANSVAGINAL OOCYTE COLLECTION

Following controlled ovarian stimulation (COS), final oocyte maturation is triggered using hCG or triptorelin. Oocyte collection is performed 35-36 hours post triggering. The procedure involves transvaginal ultradound-guided aspiration of follicles via a double lumen aspiration needle (16G, Casmed),. An interdisciplinary team is required for the procedure, including Gynaecologists, Embryologists Midwives/Nurses and Anaesthetists. It is performed in a gynaecological operating theatre, adjacent to an embryology laboratory, with the patient being sedated and under aseptic conditions and strict regulation of environmental conditions to ensure oocyte viability and patient safety.

Before the procedure The day before the procedure, the embryologist prepares culture dishes (Falcon Central Well dishes) containing bicarbonate buffered media specifically designed for oocyte culture (Fert, Origio) overlaid with mineral oil (Fertipro). The dishes are placed in a 5-7% CO2 incubator at 37oC to equilibrate overnight. Aliquots of HEPES buffered media (Flushing medium, Origio) which achieves pH regulation outside of the incubator is pre-heated to 37oC. Finally, 160 ml flasks of DPBS (phosphate buffered saline) for use in follicular flushing are placed in the theatre's incubator for pre-warming. All the embryological preparation is performed aseptically under a laminar flow hood.

The procedure utilises surgical equipment which is autoclaved and packagedd in sterile surgical cloths. All materials that come into contact with follicular fluid, such as oocyte needles, 20ml syringes (non toxic, BD) and collection tubes (14ml IVF tubes, NUNC), are IVF tested via MEA testing (mouse blastocyst survival), pre-sterilised and single use. These are stored prior to use in a 37oC warming chamber.

We use a 16G double lumen needle (Casmed, UK) which allows continuous aspiration and flushing of follicles. The needle has a length of 30 cm and echogenic markings near the tip for easy recognition under transvaginal ultrasound guidance. The length of the tubing is 60cm and includes a bung for connection to a standard test tube and separate tubing with a Luer-lock for connection to a syringe for flushing. The needle and its connections are all manufactured from high grade surgical stainless steel. The tubing is manufactured from translucent PTFE (Polytetrafluoroethylene).

All products are manufactured in accordance with quality standards ISO 9001:2008, ISO 13485 and CE marking.

Preparing for the procedure Patient Preparation Before entering the operating theatre, the anaesthesiologist confirms the patient's medical history pertinent to her imminent anaesthesia.

The patient is escorted to the operating theatre and her identity is confirmed by two persons, who sign the witnessing document. In patients with very few expected oocytes (poor responders, mild IVF or natural cycles) a transvaginal ultrasound is performed just prior to the procedure by the treating physician in order to confirm the presence and location of mature follicles. In cases of high risk for ovarian hyperstimulation syndrome, a blood sample is also taken, according to our standard clinical practice as previously described (Lainas et al., 2012, 2013, 2014). The procedure followed for the preparation of the patient is the same as that of most gynaecological surgeries. The patient is laid on the operating table in the lithotomy position and her external genitalia are washed with hibitane solution (which is considered milder than using betadine scrub) and then rinsed with saline. After performing a standard hand and arm scrub, the surgeon's assistant wears surgical gloves and opens the sterilised tool packages, including pre-warmed and sterilised tube blocks, which is placed on sterilised surgical paper towels within a heating stage. Sterilised collection tubes are placed in the heating block, for use during the procedure. If during the procedure more tubes are required the assisting nurse should aseptically place more tubes in the heating block. The patient is then covered with sterilised surgical towels on the body and legs.The probe of the ultrasound is disinfected with CIDEX for 5 minutes and then washed with copious amounts of water for injection. Following insertion of a vaginal dilator, the vagina is washed with DPBS up to the cervical os. The assistant then wears new surgical gloves and gown and covers the patient with additional sterilised surgical paper drapes The pre-sterilised oocyte needle guide is opened and it and the flushing syringes are washed with DPBS. One syringe is carefully filled with DPBS, which will be used to flush the needle and then discarded. The ultrasound probe is then aseptically placed on the patient's drapes, the needle guide is attached to it and the probe is finally connected to the ultrasound central unit. A pre-warmed 16 G double lumen oocyte collection needle is opened and the aspiration pump is set to 250 mmHG. The needle's various tubing connectors are connected to: a) the aspiration pump, b) the flushing syringe, c) the first oocyte collection tube.

The surgeon performs a standard hand and arm scrub, wears a surgical gown and surgical gloves before assuming the surgical position at the surgical table. The needle and its tubing are washed by flushing with warm DPBS before use and the first collection tube is discarded. This ensures that the entirety of the needle/tubing is filled with DPBS before puncturing the follicle. The anaesthesiologist sedates the patient and monitors her breathing and heart function throughout the procedure.

Embryological Laboratory Preparation The entire embryological procedure is performed under a laminar flow hood, with a heated stage set at 40oC in order to endure a dish temperature of 37+/-0.2 oC. The embryologist prepares central well culture dishes with HEPES media. Empty pre-heated round dishes, heat-polished glass Pasteur pipettes and an empty container for discarded follicular fluid are all placed on the heated workbench. All of the above should be clearly labelled with the patients details.

During the procedure

The physician places the oocyte collection needle into the guide and then attaches it to the transvaginal probe of the ultrasound. He then performs an ultrasound estimation of the ovaries and Douglas pouch. After he has located the follicles, he punctures the vaginal wall with the needle at a point adjacent to the first ovary and proceeds to aspirate all antral follicles. larger than (...mm).

As each follicle is aspirated, the fluid is collected in the tube and the surgeon's assistant replaces it with a new tube from the heated stage. A nurse takes the filled tube and estimates its volume based on a volumetrically marked "reference" tube. The volumetric estimation is based on a series of tubes of known volume. The tube is then quickly placed in the heating block within the embryological laboratory (via the connecting window). Tubes are placed from left to right on the heating block, with the leftmost spot being reserved for fluids from newly aspirated follicles and the rightmost positions for tubes containing flushed follicular fluid.

The embryologist takes the tube and carefully pours the contents of each tube into the dish. He then searches for the Cumulus-Oocyte Complex (COC) through his microscope. The results of this search are communicated to the physician and fall into three categories: a) COC found, b) COC not found but follicle cells present, c) COC not found and no follicle cells present. When the COC is found, the physician moves on to the next follicle, while the embryologist transfers it to the moat of the collection dish and thoroughly washes it, before moving it to the central well. If the COC is not found, the physician then proceeds to flush DPBS into the follicle via the syringe. The volume flushed should not exceed 50% of the initial volume of the follicle to avoid rupturing it, which may cause haemorrhaging of the follicle. The flushed fluid is then aspirated and the procedure is repeated as described above. This process is repeated until the COC is found or 4-5 flushes are performed. When the flushing syringe runs out of DPBS it is replaced with a new one which has been carefully and aseptically filled just prior to use (no more than 2 minutes prior to use, in order for the temperature to not drop significantly).

As the procedure continues, COCs are placed by the embryologist in the collection dish until a maximum of 10 are collected. A new dish should be used for additional COCs. Following the end of the oocyte collection, the oocytes are transferred to dishes containing Fert medium and placed in the incubator. After the embryologist has ensured that all tubes have been searched he informs the physician of the final number of oocytes retrieved. Before ending the procedure the physician scans the ovaries and Douglas pouch one last time and if excess fluid is detected, he aspirates as much as possible. Finally the physician removes the needle and probe and ensures that there is no vaginal bleeding.

Factors contributing to successful oocyte retrieval

A transvaginal oocyte retrieval is a complicated procedure with many variables that need to be accounted for in order to make it successful. Side effects from the operation can be affected by the length of the procedure, the skill of the physician and the type of needle used. The length of the procedure is primarily affected by the number of oocytes collected and the ease that these were collected. Procedures that include flushing of follicles are on average longer than those without flushing. The width of the needle (gauge) directly affects the level of vaginal bleeding and the level of pain the patient experiences due to the operation. The above variables (flushing and width of needle) have been proposed as major factors for the effectiveness of the oocyte collection, i.e. the number of oocytes retrieved.

Follicular flushing Flushing has been proposed as a method that may increase the oocyte yield due to the fact that oocytes that are not immediately retrieved from the follicle can be collected after flushing. Double lumen needles allow for flushing via the use of two channels within the needle, one for aspirating the follicles and one for flushing. However, there is controversy regarding its routine use mainly due to the fact that the procedures tend to last longer, but also due to the risk of haemorrhage and infection from flushing. Many studies have been performed over the years comparing flushing (with double lumen needles) and no flushing (with single lumen needles), with conflicting results.

A Cochrane review published in 2010, assessed the use of flushing, found no significant benefit in the use of double-lumen needles. In a recent randomised study performed in EUGONIA clinic, flushing was found to be associated with significantly higher retrieval rates compared to no flushing using a 16G Casmed double lumen needle. In addition, around 97% of oocytes collected were retrieved in the first 3 flushes and oocytes were found to have similar maturation and fertilisation rates regardless of the number of flushes required, suggesting that a small number of flushes may increase the final number of developmentally competent oocytes retrieved.

Regarding the safety of flushing, adherence to the protocol presented above, especially with regard to aseptic techniques, will minimise the risk of infection from the flushes. It should be stressed that care should be taken to avoid rupturing follicles via too vigorous flushing. The amount of DPBS flushed into the follicle should not exceed 50% of the volume of the follicle and follicles with excess vascularisation should not be flushed at all. The procedure should be performed by an experienced team to ensure safety of the patient while also minimising the length of time of the surgery.

Aspiration Needles A significant parameter when comparing both needles and retrieval techniques is the working diameter of the needle used to aspirate. This is especially true when performing oocyte retrievals with the use of follicular flushing. Double lumen needles have as a rule smaller working diameters compared to similar gauge single lumen needles. This fact should be considered when setting the negative pressure on the aspiration pump, as double-lumen needles will require significantly higher pressure in order to achieve a similar flow rate as single-lumen needles. Even similar double-lumen needles from different manufacturers can have dissimilar inner lumen diameters, significantly altering their performance, since even small changes in the diameter have a large effect on the flow-rate. Below is a comparison of the diameters of some commonly used aspiration needles. The inner diameter in the double lumen category refers to the working diameter of the inner lumen. Note the significant differences in diameters between similar gauge needles.

SINGLE LUMEN DOUBLE LUMEN 16G 16G 17G 17G 16G 16G 17G 17G OUTER INNER OUTER INNER OUTER INNER OUTER INNER WALLACE 1,7 1,24 1,42 1 1,7 1,17 1,5 0,9 GYNETICS 1,6 1,3 1,4 1 1,65 1 1,5 0,8 VITROLIFE 1,6 1,1 1,4 1 1,6 1 1,5 0,9 CASMED n/a n/a n/a n/a 1,65 0,81 n/a n/a

ELIGIBILITY:
Inclusion Criteria:

* Presence of both ovaries
* 18-40 years old
* Triggering final oocyte maturation using human chorionic gonadotrophin (hCG) or gonadotrophin releasing hormone (GnRH) agonist

Exclusion Criteria:

* One or no ovaries present
* Endometriosis
* Previous history of hemorrhage during oocyte retrieval

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be born as females and have two ovaries present
Study Population: Women undergoing IVF treatment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Oocyte recovery rate | Day of oocyte retrieval
  Number of oocytes retrieved per follicle aspirated

SECONDARY OUTCOMES:
Number of oocytes retrieved | Day of oocyte retrieval
  Number of oocytes retrieved
Oocyte maturation rate | Day of oocyte retrieval
  Number of mature (metaphase-II) oocytes per oocyte retrieved
Fertilization rate | Day 1 post oocyte retrieval
  Number of fertilized oocytes per oocyte injected/inseminated
Good quality embryos on day 2/3 | 2/3 days post oocyte retrieval
  Percentage of good quality embryos per number of fertilized oocytes
Blastocyst formation rates | Day 5 post oocyte retrieval
  Number of blastocysts formed on Day 5 per number of fertilized oocytes
Hemorrhage | Day of oocyte retrieval
  Hemorrhagic ovary during/following oocyte retrieval
Embryo cryopreservation | Day 5 post oocyte retrieval
  Number of embryos cryopreserved per total number of fertilized oocytes
Embryo utilization | Day 5 post oocyte retrieval
  Number of embryos transferred and cryopreserved per total number of fertilized oocytes
Embryos transferred | Days 2-5 post oocyte retrieval
  Number of embryos selected for transfer

CONTACTS AND LOCATIONS:
Overall Officials: Lainas, PhD, Study Director — Eugonia
Locations (1):
- Eugonia, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] von Horn K, Depenbusch M, Schultze-Mosgau A, Griesinger G. Randomized, open trial comparing a modified double-lumen needle follicular flushing system with a single-lumen aspiration needle in IVF patients with poor ovarian response. Hum Reprod. 2017 Apr 1;32(4):832-835. doi: 10.1093/humrep/dex019. PMID 28333185
- [Background] Franasiak JM. Follicular flushing: time to look elsewhere to improve in vitro fertilisation outcomes? BJOG. 2017 Jul;124(8):1197. doi: 10.1111/1471-0528.14628. No abstract available. PMID 28276189
- [Background] Roque M, Sampaio M, Geber S. Follicular flushing during oocyte retrieval: a systematic review and meta-analysis. J Assist Reprod Genet. 2012 Nov;29(11):1249-54. doi: 10.1007/s10815-012-9869-9. Epub 2012 Oct 13. PMID 23065177